CLINICAL TRIAL: NCT02956746
Title: A Phase 2 Randomized Blinded Placebo Controlled Comparison of the Safety Pharmacokinetics and Pharmacodynamics of a Single Dose of SYN023 Administered With Licensed Rabies Vaccines in Healthy Adult Subjects
Brief Title: A Comparison of the Safety, PD and PK of a Single Dose of SYN023 Administered With Licensed Rabies Vaccines
Acronym: RabiesMab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Synermore Biologics Co., Ltd. (Industry)
Collaborators: inVentiv Health Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SYN023-002
Record Dates: First submitted 2016-11-01; First posted 2016-11-07 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Human Rabies
MeSH Terms: interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Imovax, SYN023 (Experimental): Subjects will receive SYN023 and 5 doses of Imovax rabies vaccine
  Interventions: Biological: SYN023; Biological: Imovax
- Imovax, human rabies immune globulin (Active Comparator): Subjects will receive HyperRAB ST (human rabies immune globulin) and 5 doses of Imovax rabies vaccine
  Interventions: Biological: Imovax; Biological: HyperRAB ST (human rabies immune globulin)
- RabAvert, SYN023 (Experimental): Subjects will receive SYN023 and 5 doses of RabAvert rabies vaccine
  Interventions: Biological: SYN023; Biological: RabAvert
- RabAvert, human rabies immune globulin (Active Comparator): Subjects will receive HyperRAB ST (human rabies immune globulin) and 5 doses of RabAvert rabies vaccine
  Interventions: Biological: RabAvert; Biological: HyperRAB ST (human rabies immune globulin)

INTERVENTIONS:
Biological: SYN023 — The effects of SYN023 on immunogenicity of rabies vaccines Imovax and RabAvert will be compared to the effect of human rabies immune globulin.
  Arms: Imovax, SYN023; RabAvert, SYN023
Biological: Imovax — Subjects will receive SYN023 or HyperRAB ST (human rabies immune globulin) and 5 doses of Imovax rabies vaccine
  Arms: Imovax, SYN023; Imovax, human rabies immune globulin
Biological: RabAvert — Subjects will receive SYN023 or HyperRAB ST (human rabies immune globulin) and 5 doses of RabAvert rabies vaccine
  Arms: RabAvert, SYN023; RabAvert, human rabies immune globulin
Biological: HyperRAB ST (human rabies immune globulin) — The effects of SYN023 on immunogenicity of rabies vaccines Imovax and RabAvert will be compared to the effect of human rabies immune globulin.
  Arms: Imovax, human rabies immune globulin; RabAvert, human rabies immune globulin

SUMMARY:
This is single site, randomized, blinded comparison of the immunogenicity, of Imovax (RVi) and Rabavert (RVa) rabies vaccines when subjects are administered rabies immune globulin (RIG) or SYN023. Subjects will be randomized into one of four dose groups: RVi + SYN023, RVi+RIG, RVa+SYN023 and RVa+RIG. The initial dose of RVi and RVa will be co-administered with either RIG or SYN023). Rabies virus neutralizing activity (RVNA) and blood levels of SYN023 will be measured for the remainder of the trial while the rest of the five RVi and RVa doses are given. The study will last 112 days. SYN023 concentrations and anti-SYN023 antibodies will also be measured.

DETAILED DESCRIPTION:
Administered immunoglobulins directed against vaccine antigens have the potential to inhibit the immune response to a vaccine. Both vaccination and immune globulin are used together in the post exposure prophylaxis of rabies virus infection. SYN023 (a mixture of two monoclonal antibodies CTB011 and CTB012) may be used instead of human rabies immune globulin. Since there is a risk of antagonism of vaccine induced immunity by SYN023, as there is with rabies immune globulin, it is necessary to study possible interactions of these two agents that might be used concurrently. This is single site, randomized, blinded comparison of the immunogenicity, of Imovax (RVi) and Rabavert (RVa) rabies vaccines when administered concurrently with rabies immune globulin (RIG) or SYN023. Subjects will be randomized into one of four dose groups: RVi + SYN023, RVi + RIG, RVa+SYN023 and RVa + RIG. The initial dose of RVi and RVa will be co-administered with either RIG or SYN023). The remaining 4 doses of RVi and RVa will be administered intramuscularly as specified in the product labeling. Serum rabies virus neutralizing activity (RVNA) and serum concentrations of the components of of SYN023 will be measured for the remainder of the trial while the rest of the five RVi and RVa doses are given. Adverse events will be collected for the duration of the trial. The study will last 112 days. Anti-SYN023 antibodies will also be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 50 years of age, inclusive
2. Body mass index between 18 and 30 kg/m², inclusive
3. Female subjects physically capable of pregnancy (i.e., not sterilized and still menstruating or within 1 year of the last menses if menopausal) must:

   1. Agree to avoid pregnancy from 28 days prior to Study Day 0 through the duration of the study.
   2. If in a sexual relationship with a man, use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include: the use of at least two forms of contraception, including use by a partner of a barrier method (e.g., male condom with intravaginal spermicide) as one form of contraception.
4. Women of childbearing potential must have a negative serum pregnancy test within 24 hours preceding receipt of each dose.
5. Can understand and sign the informed consent document, can communicate with the investigator and provide updated contact information as needed for the duration of the study, has no current plans to move from the study area for the duration of the study, and can understand and comply with the requirements of the protocol.

Exclusion Criteria:

1. Oral temperature ≥37.5°C at screening
2. Complete blood count (CBC) and platelet count abnormal values (>5% above the upper limit of normal [ULN] or >5% below the lower limit of normal [LLN] per local laboratory parameters) at screening with exception of absolute lymphocyte count.
3. Abnormally elevated aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, alkaline phosphatase (ALP), or creatinine (Cr) values at screening (however a single test AST, ALT or ALP may be >10% above the ULN per local laboratory parameters)
4. Abnormal PT (INR) PTT
5. Abnormal screening urinalysis result that is, per the investigator, clinically significant, or a screening urine dipstick result of ≥2+ protein
6. Positive screening urine test for illicit drugs (opiates, cocaine, amphetamines methamphetamines, barbiturates, benzodiazepines, tetrahydrocannabinol, PCP, MDMA, and methadone)
7. History or evidence of autoimmune disease
8. History or evidence of any past, present, or future possible immunodeficiency state, including laboratory evidence of human immunodeficiency virus (HIV) 1 or 2 infection
9. History or evidence of chronic hepatitis
10. History or evidence of rabies infection
11. History or evidence of any other acute or chronic disease that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the drug or compromise the safety of the subject; for example a clinically relevant history of respiratory, thyroid, gastrointestinal, renal, hepatic, hematological, lymphatic, oncologic, cardiovascular, psychiatric, neurological, musculoskeletal, genitourinary, infective, inflammatory, immunological, dermatological or connective tissue disease
12. History or evidence of allergic disease or reaction, including adverse responses to therapeutic monoclonal antibodies that, in the opinion of the investigator, may compromise the safety of the subject
13. History of non-compliance that, in the opinion of the investigator, will make it unlikely that the subject will comply with the protocol
14. Previous exposure to rabies vaccine
15. Receipt of an immunoglobulin or blood product within 90 days prior to Study Day 0
16. Receipt of immunosuppressive medications other than inhaled or topical immunosuppressant drugs within 45 days prior to Study Day 0
17. Body weight greater than 90 kg.
18. History or evidence of IgA deficiency

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wyatt J David, PhD, Principal Investigator — inVentiv Health Clinical Research Services LLC
Locations (1):
- inVentiv Clinical Research Facility, 1951 NW 7th Ave. Suit 450, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McClain JB, Chuang A, Reid C, Moore SM, Tsao E. Rabies virus neutralizing activity, pharmacokinetics, and safety of the monoclonal antibody mixture SYN023 in combination with rabies vaccination: Results of a phase 2, randomized, blinded, controlled trial. Vaccine. 2021 Sep 24;39(40):5822-5830. doi: 10.1016/j.vaccine.2021.08.066. Epub 2021 Sep 3. PMID 34483020

RESULTS

PARTICIPANT FLOW:
Groups:
- Imovax, SYN023: Subjects will receive SYN023 and 5 doses of Imovax rabies vaccine
  SYN023: The effects of SYN023 on immunogenicity of rabies vaccines Imovax and RabAvert will be compared to the effect of human rabies immune globulin.
  Imovax, human rabies immune globulin: Subjects will receive HyperRAB ST (human rabies immune globulin) and 5 doses of Imovax rabies vaccine
  RabAvert, human rabies immune globulin: Subjects will receive HyperRAB ST (human rabies immune globulin) and 5 doses of RabAvert rabies vaccine
- Imovax, Human Rabies Immune Globulin: Subjects will receive HyperRAB ST (human rabies immune globulin) and 5 doses of Imovax rabies vaccine
  SYN023: The effects of SYN023 on immunogenicity of rabies vaccines Imovax and RabAvert will be compared to the effect of human rabies immune globulin.
  Imovax, human rabies immune globulin: Subjects will receive HyperRAB ST (human rabies immune globulin) and 5 doses of Imovax rabies vaccine
  RabAvert, human rabies immune globulin: Subjects will receive HyperRAB ST (human rabies immune globulin) and 5 doses of RabAvert rabies vaccine
- RabAvert, SYN023: Subjects will receive SYN023 and 5 doses of RabAvert rabies vaccine
  SYN023: The effects of SYN023 on immunogenicity of rabies vaccines Imovax and RabAvert will be compared to the effect of human rabies immune globulin.
  Imovax, human rabies immune globulin: Subjects will receive HyperRAB ST (human rabies immune globulin) and 5 doses of Imovax rabies vaccine
  RabAvert, human rabies immune globulin: Subjects will receive HyperRAB ST (human rabies immune globulin) and 5 doses of RabAvert rabies vaccine
- RabAvert, Human Rabies Immune Globulin: Subjects will receive HyperRAB ST (human rabies immune globulin) and 5 doses of RabAvert rabies vaccine
  SYN023: The effects of SYN023 on immunogenicity of rabies vaccines Imovax and RabAvert will be compared to the effect of human rabies immune globulin.
  Imovax, human rabies immune globulin: Subjects will receive HyperRAB ST (human rabies immune globulin) and 5 doses of Imovax rabies vaccine
  RabAvert, human rabies immune globulin: Subjects will receive HyperRAB ST (human rabies immune globulin) and 5 doses of RabAvert rabies vaccine
Period: Overall Study
Arm/Group | Imovax, SYN023 | Imovax, Human Rabies Immune Globulin | RabAvert, SYN023 | RabAvert, Human Rabies Immune Globulin
Started | 40 | 40 | 42 | 42
Completed | 38 | 37 | 36 | 38
Not Completed | 2 | 3 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imovax, SYN023 | Imovax, Human Rabies Immune Globulin | RabAvert, SYN023 | RabAvert, Human Rabies Immune Globulin | Total
Number analyzed (Participants) | 40 | 40 | 42 | 42 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 42 | 42 | 164
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 28 | 20 | 103
  Male | 12 | 13 | 14 | 22 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 37 | 39 | 40 | 153
  Not Hispanic or Latino | 3 | 3 | 3 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 42 | 42 | 164
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.41 (2.87) | 25.74 (2.96) | 24.92 (2.66) | 24.39 (3.14) | 24.86 (2.93)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Rabies Virus Neutralizing Activity
Description: Inhibitory activity of serum in standard rabies virus inhibition test (RFFIT: Rapid Fluorescent Foci Inhibition Test) assessed as serum RVNA ≥ 0.5 IU/mL. RFFIT is a serum neutralization (inhibition) test, which means it measures the ability of rabies specific antibodies to neutralize rabies virus and prevent the virus from infecting cells. These antibodies are called rabies virus neutralizing antibodies (RVNA).
Time Frame: 112 days
Population: Per-Protocol Population (subject with complete RVNA data).
Measure: Number; unit: percentage of participants
Arm/Group | Imovax, SYN023 | Imovax, Human Rabies Immune Globulin | RabAvert, SYN023 | RabAvert, Human Rabies Immune Globulin
Number analyzed (Participants) | 35 | 35 | 34 | 36
percentage of participants | 94.3 | 97.1 | 97.1 | 100
Statistical Analysis 1: Comparison: Imovax, SYN023 vs Imovax, Human Rabies Immune Globulin vs RabAvert, SYN023 vs RabAvert, Human Rabies Immune Globulin; Test type: Other; p = 0.4187, ANOVA — threshold for significance p-values < 0.05

2. Secondary Outcome: Percentage of Participants With Adverse Event Incidence of SYN023 Compared to HRIG in RabAvert and Imovax Reciptients
Description: Electrocardiograms are performed to monitor subject safety. Laboratory evaluations for subject safety (adverse events) are serum chemistry evaluations, blood urea nitrogen, creatinine, bilirubin, alanine amino transferase, aspartate amino transferase, creatine phosphokinase, troponin, potassium, sodium, bicarbonate, calcium, complete blood count, platelet count, differential count, PT(prothrombin time, international normalized ratio) and PTT (partial prothrombin time and urinalyses for monitoring of safety. Additional laboratory tests may be required for evaluation of specific adverse events such as anaphylaxis and immune complex diseases. Adverse events and serious adverse events will be analyzed. A comparison of adverse event incidence between the four treatment groups will be performed.
Time Frame: 42 days
Measure: Number; unit: percentage of participants
Arm/Group | Imovax, SYN023 | Imovax, Human Rabies Immune Globulin | RabAvert, SYN023 | RabAvert, Human Rabies Immune Globulin
Number analyzed (Participants) | 40 | 40 | 42 | 42
percentage of participants
  Unsolicited AEs | 60 | 50 | 73.8 | 59.5
  Solicited AEs | 15 | 47.5 | 28.6 | 40.5

3. Secondary Outcome: Percentage of Participants With Immunogenicity: Anti-CTB012 Antibodies Positive
Description: Measurement of the development of anti-CTB012 antibodies (a component of anti-SYN023 antibodies) in participants which will be analyzed on a continuous scale as a categorical variable by treatment assignment, with descriptive statistics.
Time Frame: 112 days
Population: Subjects at least 1 initial anti-SYN023 assay results
Measure: Number; unit: percentage of participants
Arm/Group | Imovax, SYN023 | Imovax, Human Rabies Immune Globulin | RabAvert, SYN023 | RabAvert, Human Rabies Immune Globulin
Number analyzed (Participants) | 40 | 30 | 42 | 31
percentage of participants | 5.3 | 0 | 0 | 3.6

4. Secondary Outcome: Percentage of Participants With Immunogenicity: Anti-CTB011 Antibodies Positive
Description: Measurement of the development of anti-CTB011 antibodies (a component of anti-SYN023 antibodies) in participants which will be analyzed on a continuous scale as a categorical variable by treatment assignment, with descriptive statistics.
Time Frame: 112 days
Population: Subjects at least 1 initial anti-SYN023 assay results
Measure: Number; unit: percentage of subjects
Arm/Group | Imovax, SYN023 | Imovax, Human Rabies Immune Globulin | RabAvert, SYN023 | RabAvert, Human Rabies Immune Globulin
Number analyzed (Participants) | 40 | 30 | 42 | 31
percentage of subjects | 36.8 | 28.6 | 31.4 | 21.4

5. Secondary Outcome: SYN023 Monoclonal Antibody Areas Under the Curve (AUC0-last, AUC0-inf) for CTB011 and CTB012)
Description: The area under the time concentration curve for SYN023 mAb components CTB011 and CTB012 will be estimated at Day 0 ( pre-dose), Day 1, Day 3, Day 7, Day 14, Day 28, Day 35, Day 42, and Day 84 post-dose, using non compartmental analysis.
Time Frame: 84 days
Population: Per-Protocol Population (subjects who received all scheduled doses of a study treatment and remained on study for at least 28 days without major protocol violation)
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Imovax, SYN023 | RabAvert, SYN023
Number analyzed (Participants) | 38 | 37
day*ng/mL
  AUC0-t for CTB-011 | 17549.49 (8300.05) | 17318.95 (7488.84)
  AUC0-inf for CTB-011 | 20604.56 (8904.60) | 20924.6 (7041.56)
  AUC0-t for CTB-012 | 22896.71 (113653.68) | 23617.93 (10768.7)
  AUC0-inf for CTB-012 | 30943.29 (11230.39) | 32495.98 (11892.98)

6. Secondary Outcome: Time to Maximum Concentration Tmax of CTB011 and CTB012
Description: Interval from time 0 to maximum measured concentration of CTB011 and CTB012 (SYN023 components) at Day 0 ( pre-dose), Day 1, Day 3, Day 7, Day 14, Day 28, Day 35, Day 42, and Day 84 post-dose, using non compartmental analysis.
Time Frame: 84 days
Population: Per-Protocol Population (subjects who received all scheduled doses of a study treatment and remained on study for at least 28 days without major protocol violation). No detectable and quantifiable levels of CTB011 and CTB012 were observed in human rabies immune globulin groups, so no PK or statistical analysis was planned.
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Imovax, SYN023 | RabAvert, SYN023
Number analyzed (Participants) | 38 | 37
day
  Tmax for CTB-011 | 6.655 (5.957) | 6.686 (4.741)
  Tmax for CTB-012 | 6.892 (6.316) | 6.932 (4.417)

7. Secondary Outcome: Maximum Serum Concentration Cmax
Description: Maximum concentration of of CTB011 and CTB012 at Day 0 ( pre-dose), Day 1, Day 3, Day 7, Day 14, Day 28, Day 35, Day 42, and Day 84 post-dose, using non compartmental analysis.
Time Frame: 84 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Imovax, SYN023 | RabAvert, SYN023
Number analyzed (Participants) | 38 | 37
ng/mL
  Cmax for CTB-011 | 686 (292) | 610 (240)
  Cmax for CTB-012 | 959 (449) | 879 (400)

8. Secondary Outcome: Serum Clearance Rate (Clp) of CTB011 and CTB012
Description: Calculated serum clearance rates for CTB011 and CTB012 at Day 0 ( pre-dose), Day 1, Day 3, Day 7, Day 14, Day 28, Day 35, Day 42, and Day 84 post-dose, using non compartmental analysis.
Time Frame: 84 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | Imovax, SYN023 | RabAvert, SYN023
Number analyzed (Participants) | 38 | 37
L/day
  clearance rates for CTB011 | 1.18 (0.62) | 1.14 (0.59)
  clearance rates for CTB012 | 0.74 (0.29) | 0.77 (0.46)

9. Secondary Outcome: Serum Half Lives of CTB011 and CTB012
Description: The time in hours to reduce the serum concnetration of CTB011 and CTB012 to 50% of the maximum serum concentration at Day 0 ( pre-dose), Day 1, Day 3, Day 7, Day 14, Day 28, Day 35, Day 42, and Day 84 post-dose, using non compartmental analysis.
Time Frame: 84 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Imovax, SYN023 | RabAvert, SYN023
Number analyzed (Participants) | 38 | 37
day
  t1/2 for CTB-011 | 19.19 (6.64) | 22.12 (5.18)
  t1/2 for CTB-012 | 20.76 (8.73) | 22.86 (8.7)

ADVERSE EVENTS:
Time Frame: 112 days
Arm/Group | Imovax, Human Rabies Immune Globulin | RabAvert, Human Rabies Immune Globulin | Imovax, SYN023 | RabAvert, SYN023
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/42 | 0/40 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42 | 0/40 | 1/42
Other Adverse Events (participants affected / at risk) | 20/40 | 25/42 | 24/40 | 31/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imovax, Human Rabies Immune Globulin (N=40) | RabAvert, Human Rabies Immune Globulin (N=42) | Imovax, SYN023 (N=40) | RabAvert, SYN023 (N=42)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imovax, Human Rabies Immune Globulin (N=40) | RabAvert, Human Rabies Immune Globulin (N=42) | Imovax, SYN023 (N=40) | RabAvert, SYN023 (N=42)
Injection site pain (General disorders) | 7 (7) | 6 (7) | 11 (11) | 20 (21)
Influenza like illness (General disorders) | 1 (1) | 3 (4) | 0 (0) | 3 (3)
Vessel puncture site bruise (General disorders) | 2 (2) | 2 (3) | 1 (1) | 2 (2)
Injection site erythema (General disorders) | 3 (4) | 0 (0) | 1 (1) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
Injection site bruising (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Energy increased (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red blood cells urine positive (Investigations) | 1 (1) | 5 (6) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 6 (7)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Muscle contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT02956746/SAP_000.pdf
  • Study Protocol (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT02956746/Prot_001.pdf